CLINICAL TRIAL: NCT04873622
Title: Addressing Stress Responses on the Frontline-Further Development of RESTORE (Recovering From Extreme Stressors Through Online Resources and E-health)
Brief Title: Further Development and Initial Testing of RESTORE in Frontline Workers
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Department of Defence (Unknown); University Health Network Foundation (Unknown)
Responsible Party: Principal Investigator, Kathryn Trottier, Psychologist and Clinical Program Lead, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB# 20-5546-1
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Mental Health; PTSD; Anxiety; Depressive Symptoms
Keywords: eHealth intervention; COVID-19; mental health
MeSH Terms: conditions — Psychological Well-Being; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RESTORE intervention (Experimental): Participants who screen eligible and consent will receive RESTORE with guidance.
  Interventions: Behavioral: RESTORE: Recovering from Extreme Stressors Through Online Resources and E-health

INTERVENTIONS:
Behavioral: RESTORE: Recovering from Extreme Stressors Through Online Resources and E-health — RESTORE (www.restoreonline.ca) includes eight e-modules anticipated to be approximately 30-40 minutes each in length and intended to be completed over 4-8 weeks. The modules address cognitive and behavioural factors posited to cause and maintain psychological distress related to the COVID-19 pandemic. These include cognitions about the cause and meaning of stressors related to the pandemic, including self-blame, other blame and hindsight bias, as well as problematic beliefs related to safety, trust, and control. The modules also address the importance of: (1) expressing emotions that are natural to the events of the pandemic (e.g., sadness in the face of loss), (2) working through, rather than avoiding, thoughts, feelings and grief related to the pandemic, and (3) utilizing social supports. The modules consist of written materials, brief videos, and practice assignments delivered through the platform. RESTORE includes guidance via direct messaging and/or brief telephone calls.

SUMMARY:
There is considerable need for psychological intervention targeting stressor-related mental health symptoms related to COVID-19. The investigators have developed an online self-directed transdiagnostic intervention to address this need called RESTORE: Recovering from Extreme Stressors Through Online Resources and E-health. The specific aims of this project are to refine and investigate the feasibility, initial safety, and efficacy of RESTORE for addressing mental health symptoms in first responders, health care workers (HCW), and Canadian Armed Forces members exposed to COVID-19-related traumatic or extreme stressors.

DETAILED DESCRIPTION:
This uncontrolled pilot interventional study will examine the feasibility and preliminary efficacy of RESTORE. RESTORE is a guided self-directed online intervention to improve anxiety, depression, and posttraumatic stress disorder (PTSD) in individuals exposed to COVID-19 related traumatic or extreme stressors. RESTORE is based on evidence-based psychotherapies and has been designed to overcome many of the barriers associated with accessing evidence-based psychotherapies. The intervention will be iteratively refined over the course of the study. The guidance methods will also be refined and manualized over the course of the study

The primary hypotheses are that RESTORE will be safe, feasible, and desirable to participants, and will lead to improvements in mental health symptom severity from baseline to post-intervention. Secondary hypotheses are that RESTORE will lead to significant improvements in perceived health, quality of life, and functioning from baseline to post-intervention. Participants will be assessed at baseline, pre-intervention, during the intervention (after module 4), immediately after the intervention, and 1 month after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Canadian healthcare worker, first responder, or military member
* Experienced a traumatic or extremely stressful situation in the course of work related to COVID-19
* ≥ 18 years of age
* Scores at above clinical threshold, as defined by the investigators, on at least one of: Patient Health Questionnaire-9 ([PHQ-9] score ≥ 10), Generalized Anxiety Disorder Scale-7 ([GAD-7] score ≥ 10), and/or Posttraumatic Stress Disorder Scale-5 ([PCL-5] score ≥ 33)
* Access to a computer or a tablet with high speed internet access, be able to clearly see the screen of a computer or tablet, and be fluent in English
* Ability to provide consent

Exclusion Criteria:

* Elevated risk of suicide
* Currently enrolled in another intervention or treatment (e.g., cognitive behavioural therapy) for stress responses related to the COVID-19 pandemic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Change in self-reported Post Traumatic Stress Disorder (PTSD) symptoms | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  The PTSD Checklist-5 (PCL-5); Weathers, Litz, Keane, Palemeri, Marx, & Schnurr, 2013) weekly version will provide a measure of change in self-reported PTSD symptoms over the course of intervention. Items are rated from 0 (not at all) to 4 (extremely). Items are summed to create a total score ranging from 0 to 80. A cutoff score of ≥ 33 can be used for screening for PTSD diagnosis (Weathers et al, 2013).
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  A brief clinical measure to assess anxiety severity. Each item is rated on a 4-point scale from 0 (not at all) to 3 (nearly every day). A symptom severity score is calculated based on the sum of the 7 items, with scores ranging from 0 to 21. GAD-7 scores of 10 and 15 are the cut-off points for moderate and severe anxiety, respectively (Spitzer et., 2006).
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  A self-report measure of depression symptoms. Each of the 9 items is rated on a 4-point scale, ranging from 0 (not at all) to 3 (nearly every day). Items are summed to produce a total severity score ranging from 0 to 27, with higher scores indicating greater symptom severity. PHQ-9 scores ≥ 10 are considered indicative of moderate levels of depression (Manea et al., 2011).

SECONDARY OUTCOMES:
Change in Perceived Health, Functioning, and Quality of Life (QOL) | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  Single items will be used to measure perceived health, work functioning, and quality of life over the past month. Each item is rated on a 5-point scale, ranging from 1 (not at all satisfied/poor) to 5 (extremely satisfied/excellent).
Change in Trauma-Related Guilt Inventory (TRGI) | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  The TRGI is a 32-item self-report questionnaire designed to measure guilt experienced as a result of surviving a traumatic event. The inventory includes three scales: guilt cognitions, distress, and global guilt scales.
Change in Adapted Brief Grief Questionnaire | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  The Adapted Brief Grief Questionnaire is a 5-item self-report measure for screening for complicated grief (Shear et al., 2006). The items deal with difficulty accepting the death, interference in current life, troubling thoughts related to the death, avoidance of reminders of the loss, and feeling distant from others. Each item is scored from 0 to 2 (0 = not at all, 1 = somewhat, 2 = a lot).
Change in Perceived emotional social support | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  Perceived Emotional Social Support is a single item measure of emotional of social support received in the past week from family and friends (Stappenbeck et al., 2015). The item is rated on a 5-point Likert scale, with responses ranging from 1 (strongly disagree) to 5 (strongly agree).
Change in Adapted Expressions of Moral Injury Scale | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  The Adapted Expressions of Moral Injury Scale is an investigator-adapted version of the Expressions of Moral Injury Scale (EMES). The EMES is a brief measure assessing emotions, beliefs, and behaviours associated with moral injury (Koenig, Mantri, Wang, & Lawson, 2020). Each of the 11 items is rated on a 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Change in Mental Health Seeking Attitudes/Intention Scale | Baseline, pre-intervention; during the intervention (after module 4); immediately after the intervention; 1-month follow-up
  The Mental Health Seeking Attitudes/Intention Scale is an adapted 3-item measure to assess attitudes toward seeking help from a mental health professional (Hammer, Parent, & Spiker, 2018). Each of the items is rated on a 7-point scale, ranging from 1 (definitely false) to 7 (definitely true).

OTHER OUTCOMES:
Qualitative interviews | Immediately after the intervention
  Qualitative interviews will be conducted post-intervention to further assess acceptability and to improve RESTORE content and presentation.
Feasibility of recruitment | After enrolment
  Feasibility of recruitment measured by percentage of screened individuals who are eligible and percentage of those who screen eligible who are subsequently enrolled.
Intervention adherence | Immediately after the intervention
  Adherence to the intervention measured by mean number of completed modules and drop out rate.
Intervention engagement | Immediately after the intervention
  Engagement will be measured by mean number of platform log-ins, mean number of module entries and mean number of practice assignment entries.
Client Satisfaction Questionnaire | Immediately after the intervention
  At the end of the intervention, participants will complete the Client Satisfaction Questionnaire (Attkisson & Zwick, 1982), which measures client satisfaction with the intervention they received. This short questionnaire consists of 6 items, and each item is rated on a 4-point scale with varying response alternatives (1=poor/no, definitely not/quite dissatisfied to 4=excellent/yes, definitely/very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Trottier, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- UHN - Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammer JH, Parent MC, Spiker DA. Mental Help Seeking Attitudes Scale (MHSAS): Development, reliability, validity, and comparison with the ATSPPH-SF and IASMHS-PO. J Couns Psychol. 2018 Jan;65(1):74-85. doi: 10.1037/cou0000248. PMID 29355346
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kubany, E. S., Haynes, S. N., Abueg, F., Manke, F. P., Brennan, J. M., Stahura, C. (1996). Development and Validation of the Trauma-Related Guilt Inventory (TRGI). Psychological Assessment, 8, 428-444. https://doi.org/10.1037/1040-3590.8.4.428
- [Background] Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. CMAJ. 2012 Feb 21;184(3):E191-6. doi: 10.1503/cmaj.110829. Epub 2011 Dec 19. PMID 22184363
- [Background] Mantri S, Lawson JM, Wang Z, Koenig HG. Identifying Moral Injury in Healthcare Professionals: The Moral Injury Symptom Scale-HP. J Relig Health. 2020 Oct;59(5):2323-2340. doi: 10.1007/s10943-020-01065-w. PMID 32681398
- [Background] Shear KM, Jackson CT, Essock SM, Donahue SA, Felton CJ. Screening for complicated grief among Project Liberty service recipients 18 months after September 11, 2001. Psychiatr Serv. 2006 Sep;57(9):1291-7. doi: 10.1176/ps.2006.57.9.1291. PMID 16968758
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stappenbeck CA, Hassija CM, Zimmerman L, Kaysen D. Sexual assault related distress and drinking: the influence of daily reports of social support and coping control. Addict Behav. 2015 Mar;42:108-13. doi: 10.1016/j.addbeh.2014.11.013. Epub 2014 Nov 20. PMID 25437266
- [Background] The World Health Organization Quality of Life Assessment (WHOQOL): development and general psychometric properties. Soc Sci Med. 1998 Jun;46(12):1569-85. doi: 10.1016/s0277-9536(98)00009-4. PMID 9672396
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., et al. (2013). The PTSD Checklist for DSM-5 (PCL-5). Retrieved from http://www.ptsd.va.gov/professional/assessment/adult-sr/
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Derived] Trottier K, Monson CM, Kaysen D, Wagner AC, Liebman RE, Abbey SE. Initial findings on RESTORE for healthcare workers: an internet-delivered intervention for COVID-19-related mental health symptoms. Transl Psychiatry. 2022 Jun 1;12(1):222. doi: 10.1038/s41398-022-01965-3. PMID 35650179